CLINICAL TRIAL: NCT06559059
Title: Evaluating the Implementation of a Comprehensive Multilevel Virtual Oncology Program Among Veterans Diagnosed With Lung, Colorectal, Prostate, and Breast Cancers in the US Department of Veterans Affairs
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 22-01448; 5P50CA271358 (NIH)
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer Diagnosis; Colorectal Cancer (Diagnosis); Prostate Cancer Diagnosis; Breast Cancer Diagnosis
MeSH Terms: conditions — Colorectal Neoplasms; Disease; Breast Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Veterans: Veterans aged 18 years or older newly diagnosed with lung, colorectal, prostate or breast cancer. Patient records will be observed of Veterans with a new cancer diagnosis of the lung, prostate, breast, or colon and a telehealth visit utilizing the VA National TeleOncology Service (NTO).
- VA health care providers and staff members: VA health care providers and staff members participating in cancer care at NTO program medical centers, including physicians, nurse practitioners, physicians' assistants and nurses.

SUMMARY:
The objective of the pragmatic trial to test the effectiveness of an existing, ongoing clinical service, the VA National TeleOncology program (NTO), a multilevel telehealth population health management program. The primary aims are to study the intervention and determine its effectiveness on telehealth engagement, clinical quality, and healthcare cost outcomes across personal characteristics.

DETAILED DESCRIPTION:
Study staff will use the Veterans Health Information Systems and Technology Architecture (VistA), the VA health information technology system, to identify eligible patients at VA sites based on listed inclusion and exclusion criteria. Patient records will be observed of Veterans with a new cancer diagnosis of the lung, prostate, breast, or colon and a telehealth visit utilizing the VA National TeleOncology Service (NTO).

ELIGIBILITY:
Patients Inclusion Criteria:

1. A Veteran
2. Aged 18 years or older
3. Newly diagnosed with lung, prostate, breast, or colon cancer within 3 months of telemedicine visit
4. Engaged in an oncology visit during the 36-month analysis period at a Veterans Affairs Medical Center (VAMC) location.

VAMC Providers and Staff Inclusion Criteria:

1. Provider or staff member at one of the VAMC locations including physicians, nurse practitioners, physicians' assistants, and nurses caring for Veterans
2. Providers or staff members having helped provide care for at least 5 Veterans with cancer in the previous 6 months at a VAMC location

Patients Exclusion Criteria:

1. Veterans who have not seen any providers in the VA within the past year
2. Patients previously diagnosed with lung, prostate, breast, or colon cancer
3. Pregnant patients

VAMC Providers and Staff Exclusion Criteria:

1. Providers or staff members who do not help treat Veterans with specified cancers in oncology at the VA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans aged 18 years or older newly diagnosed with lung, colorectal, prostate or breast cancer.
  VA health care providers and staff members participating in cancer care at NTO program medical centers, including physicians, nurse practitioners, physicians' assistants and nurses.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of raw telehealth visits | Post-NTO implementation (up to 3 months)
  Telehealth utilization among Veterans with cancer will be measured through raw telehealth visit counts.
Fraction of patients engaging in at least one telehealth visit | Post-NTO implementation (up to 3 months)
  Telehealth utilization among Veterans with cancer will be measured by fraction of patients engaging in at least one telehealth visit.

SECONDARY OUTCOMES:
Change in provider level Quality Oncology Practice Initiative (QOPI) score | Pre-implementation, post-NTO implementation (up to 3 months)
  The quality of care of the intervention will be evaluating utilizing the American Society of Clinical Oncology Practice Initiative (QOPI) performance measures. The scale consists of 26 performance measures assessed at the patient, provider, and facility levels. Each cancer care provider will have his or her patient QOPI measures aggregated together for a provider level QOPI score. Our primary interest is the difference in QOPI score by intervention condition, as estimated by the fixed-effect coefficient for the intervention indicator variable. Scores of 75% or more indicate the standard is met, scores less than 75% indicate the standards have not been met. An increase in the QOPI score indicates improvement.
Time of consultation to time of first appointment | Pre-implementation, post-NTO implementation (up to 3 months)
  Time to care will be measured through time of consultation to time of first appointment.
Time of consultation to time of first treatment | Pre-implementation, post-NTO implementation (up to 3 months)
  Time to care will be measured through time of consultation to time of first treatment.
Average total cost for cancer diagnosis, treatment and downstream HealthCare utilization | Post-NTO implementation (up to 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Danil Makarov, MD, MHS, Principal Investigator — NYU Langone Health
Locations (5):
- United States (5):
  - VA New York Harbor Healthcare System - Brooklyn, Brooklyn, New York
  - VA New York Harbor Healthcare System - St. Albans Community Living Center, Jamaica, New York
  - VA New York Harbor Health Care System - Manhattan, New York, New York
  - VA New York Harbor Healthcare System - Harlem Community Center, New York, New York
  - VA New York Harbor Healthcare System - Staten Island Community Clinic, Staten Island, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data for survey and interview participants who have been consented and signed Health Insurance Portability and Accountability Act (HIPAA) waivers will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Per Veterans Health Administration (VHA) policy, the deidentified national data is unable to be shared. Requests may be directed to: janeth.juarezpadilla@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to janeth.juarezpadilla@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.